CLINICAL TRIAL: NCT06626815
Title: The Effect of Different Kangaroo Positions Given During Heel Lance Procedure on Newborns Pain, Comfort, and Physiological Parameters
Brief Title: The Effect of Different Kangaroo Positions on Newborns During Heel Lancing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/13-03
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Heel Lancing; Heel Lance Procedures; Kangaroo Mother Care; Skin to Skin Contact
Keywords: reverse kangaroo mother care; lateral kangaroo mother care; kangaroo positions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classic kangaroo position group (control group) (No Intervention)
- Lateral kangaroo position group (Experimental)
  Interventions: Behavioral: Lateral Kangaroo Position
- Reverse kangaroo position group (Experimental)
  Interventions: Behavioral: Reverse Kangaroo Position

INTERVENTIONS:
Behavioral: Lateral Kangaroo Position — Newborns in the lateral kangaroo position group will be positioned diagonally on their mothers chests, with their heads placed between the mothers breast and collarbone.
  Arms: Lateral kangaroo position group
Behavioral: Reverse Kangaroo Position — Newborns in the reverse kangaroo position group will be positioned vertically with their backs in contact with the mothers chest.
  Arms: Reverse kangaroo position group

SUMMARY:
Newborn screenings are crucial preventive health services within public health programs worldwide. In our country, as part of this program, heel blood is taken from newborns between the 48th and 72nd hours after birth, which causes pain and discomfort in newborns. Non-pharmacological methods are frequently utilized to relieve the pain caused by heel blood collection in newborns and to improve comfort during the procedure. One of these methods is kangaroo care, also known as skin-to-skin contact. Kangaroo care involves placing the baby in direct skin contact with the mother, which helps regulate the babys body temperature, calm the baby, and fosters bonding between mother and baby. This method, also described as human incubator care requires no special skills, is cost-effective, and is reported to have significant benefits in reducing procedural pain. In the literature, apart from the classic kangaroo position where the babys chest touches the mothers chest, there are studies describing alternative positions such as side kangaroo (kangaroo-supported diagonal flexion) and reverse kangaroo (supine kangaroo). The side kangaroo position differs from the classic kangaroo care in that the baby is held crosswise with its neck supported by the mother, allowing mother and baby to face each other. The reverse kangaroo position is a modified version of the classic kangaroo position, where the baby, wearing only a diaper, is placed upright with its back in contact with the mothers bare chest. Skin-to-skin contact during kangaroo care has a calming effect, reducing both physiological and behavioral pain responses in the baby. Therefore, it is thought that different kangaroo positions, which maintain skin-to-skin contact between the baby and the mother, may affect pain, comfort, physiological parameters, and crying durations during the heel blood collection procedure. Additionally, in cases where the classic kangaroo position cannot be used, these positions may serve as alternative methods. Upon reviewing national and international literature, no studies were found comparing the effectiveness of different kangaroo positions during heel blood collection in term newborns. Thus, this study aims to compare the effects of classic kangaroo, side kangaroo, and reverse kangaroo positions on pain, comfort, and physiological parameters (heart rate, oxygen saturation) in term newborns. Secondary outcomes of the study include evaluating the crying duration of newborns and the procedure duration for heel blood collection.

ELIGIBILITY:
Inclusion Criteria

* Born between 38-42 weeks of gestation
* Delivered via cesarean section
* Birth weight of 2500 grams or more
* APGAR score over 6 at 5 minutes
* Fed at least one hour prior to the procedure
* Postnatal age of 48-72 hours
* Successful heel blood collection performed in a single attempt
* No invasive procedures performed after birth, except for vitamin K and Hepatitis B vaccination
* Term newborns whose mothers have agreed to participate in the study

Exclusion Criteria for the Study

* Genetic or congenital anomalies
* Neurological, cardiological, or metabolic diseases
* Requirement for respiratory support
* Use of analgesics, sedatives, antiepileptics, or muscle relaxants within 24 hours prior to the procedure
* Mothers with physical barriers preventing kangaroo care
* Newborns whose mothers cannot communicate or do not speak Turkish

Ages: 48 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale - NIPS | Before the procedure (-5 minutes), during the procedure (0 minutes), and after the procedure (1 and 5 minutes)
  It evaluates the baby's pain through six criteria: facial expression, crying, breathing pattern, arms, legs, and alertness. Five of these criteria are scored as either 0 or 1, while crying is scored from 0 to 2, ranging from good to poor. According to this scale, a newborn's pain is assessed on a total score where the highest score is 7 and the lowest is 0. If the pain score is between 0 and 2, it is considered no pain, and no intervention is needed. If the pain score is between 3 and 4, it is assessed as moderate pain, non-pharmacological interventions are applied, and pain is re-evaluated after 30 minutes. If the pain score is above 4, non-pharmacological interventions are conducted, possibly alongside pharmacological treatments, and pain is re-evaluated after 30 minutes.
Newborn Comfort Behavior Scale - COMFORTneo | Before the procedure (-5 minutes), during the procedure (0 minutes), and after the procedure (1 and 5 minutes)
  The Newborn Comfort Behavior Scale is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. For newborns receiving mechanical ventilator support, the "Respiratory Response" parameter is evaluated, while for those not on mechanical ventilator support, the "Crying" item is assessed.
Heart rate | Before the procedure (-5 minutes), during the procedure (0 minutes), and after the procedure (1 and 5 minutes)
  It will be measured using a pulse oximeter.
Oxygen saturation | Before the procedure (-5 minutes), during the procedure (0 minutes), and after the procedure (1 and 5 minutes)
  It will be measured using a pulse oximeter.
Duration of crying | From the heel lancing until the end of the blood collection procedure
  It will be measured in seconds.
Time taken for heel blood collection | From the heel lancing until the end of the blood collection procedure
  It will be measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Aközlü, Study Director — Istanbul University - Cerrahpasa; Seda Çağlar, PhD, Study Chair — Istanbul University - Cerrahpasa; Tuğba Erener Ercan, PhD, Principal Investigator — Maltepe University
Locations (1):
- Istanbul University-Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No